CLINICAL TRIAL: NCT01160523
Title: Promoting Consistent Shoe Use Among Children At High Risk for Podoconiosis
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910142; 10-HG-N142
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-04-14

CONDITIONS: Podoconiosis; Non-Filarial Elephantiasis
Keywords: Podoconiosis; Genetic Education; Primary Prevention; Ethiopa; Youth
MeSH Terms: conditions — Elephantiasis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background: Podoconiosis is a debilitating condition affecting one million people in Ethiopia. Podoconiosis is preventable if those at genetically high risk consistently protected their feet from exposure to silica nanoparticles present in clay soil. Despite the efforts of a local Non-Government Organization (NGO) the Mossy Foot Prevention & Treatment Association (MFTPA) to distribute shoes to podoconiosis patients and their children, use of footwear is intermittent. This protocol proposes a collaboration among faculty from NHGRI, Addis Ababa University, and the MFTPA to develop and test intervention approaches that have the potential to be sustained by the community, to motivate children from families affected by podoconiosis to consistently wear shoes.

Objective: The three primary aims are to: (1) use qualitative assessment strategies to explore factors influencing shoe use among high-risk children; (2) use these findings to develop culturally-tailored intervention modules; and (3) evaluate in a randomized trial the individual and joint effects of the intervention modules in encouraging high-risk children to consistently wear shoes.

Population: Children (ages 9 -15) from families affected by podoconiosis who are participating in shoe distributions in one of 13 communities in the Wolaita zone of Ethiopia served by MFTPA.

Methods: Guided by the PRECEDE-PROCEED approach to planning, implementing and evaluating public health programs, a two-phase study is proposed.

Phase 1 will employ qualitative methods including participant observation, extended case studies, key-informant interviews and focus group discussions in a sample of 4 communities to gain understanding of the factors that influence shoe wear among high-risk children. Informed by these results, content for two modules (an enhanced education module and a role model support module) will be developed with the aim to motivate consistent use of footwear.

Phase 2 will evaluate the individual and joint effectiveness of the two intervention modules in a randomized 2 x 2 factorial design with communities assigned randomly to one of 4 intervention conditions: (GP1) no enhanced health education and no role model support (usual care), (GP2) enhanced health education without role model support, (GP3) no enhanced health education with role model support, and (GP4) enhanced health education and role model support. All children receive shoes. Children will be surveyed at baseline, 3-5 days after shoe distribution, and again, 3- and 6- months post baseline.

Outcomes: The primary outcome is a composite of direct observation of shoe use, self-reported shoe use, and baseline-to-follow-up changes in the children s foot appearance based on a visual foot exam.

...

DETAILED DESCRIPTION:
Background: Podoconiosis is a debilitating condition affecting one million people in Ethiopia. Podoconiosis is preventable if those at genetically high risk consistently protected their feet from exposure to silica nanoparticles present in clay soil. Despite the efforts of a local Non-Government Organization (NGO) the Mossy Foot Prevention & Treatment Association (MFTPA) to distribute shoes to podoconiosis patients and their children, use of footwear is intermittent. This protocol proposes a collaboration among faculty from NHGRI, Addis Ababa University, and the MFTPA to develop and test intervention approaches that have the potential to be sustained by the community, to motivate children from families affected by podoconiosis to consistently wear shoes.

Objective: The three primary aims are to: (1) use qualitative assessment strategies to explore factors influencing shoe use among high-risk children; (2) use these findings to develop culturally-tailored intervention modules; and (3) evaluate in a randomized trial the individual and joint effects of the intervention modules in encouraging high-risk children to consistently wear shoes.

Population: Children (ages 9 -15) from families affected by podoconiosis who are participating in shoe distributions in one of 13 communities in the Wolaita zone of Ethiopia served by MFTPA.

Methods: Guided by the PRECEDE-PROCEED approach to planning, implementing and evaluating public health programs, a two-phase study is proposed.

Phase 1 will employ qualitative methods including participant observation, extended case studies, key-informant interviews and focus group discussions in a sample of 4 communities to gain understanding of the factors that influence shoe wear among high-risk children. Informed by these results, content for two modules (an enhanced education module and a role model support module) will be developed with the aim to motivate consistent use of footwear.

Phase 2 will evaluate the individual and joint effectiveness of the two intervention modules in a randomized 2 x 2 factorial design with communities assigned randomly to one of 4 intervention conditions: (GP1) no enhanced health education and no role model support (usual care), (GP2) enhanced health education without role model support, (GP3) no enhanced health education with role model support, and (GP4) enhanced health education and role model support. All children receive shoes. Children will be surveyed at baseline, 3-5 days after shoe distribution, and again, 3- and 6- months post baseline.

Outcomes: The primary outcome is a composite of direct observation of shoe use, self-reported shoe use, and baseline-to-follow-up changes in the children s foot appearance based on a visual foot exam.

ELIGIBILITY:
* INCLUSION CRITERIA:

Children 9-15 years of age who have been identified to participate in the MFTPA shoe distribution.

EXCLUSION CRITERIA:

* Children younger than 9 or older than 15
* Children who show clinical evidence of podoconiosis or have confirmed diagnosis of another pathology that might affect participation in study activities (for example tuberculosis)
* Children for whom we are unable to gain parental permission.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2106 (Actual)
Dates: Start 2010-06-14; Study Completion 2016-04-14

CONTACTS AND LOCATIONS:
Overall Officials: Vence L Bonham, J.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- School of Public Health Addis Ababa University, Addis Ababa, Ethiopia

REFERENCES:
- [Background] Abebe T, Aase A. Children, AIDS and the politics of orphan care in Ethiopia: the extended family revisited. Soc Sci Med. 2007 May;64(10):2058-69. doi: 10.1016/j.socscimed.2007.02.004. Epub 2007 Mar 26. PMID 17379371
- [Background] Ayaya SO, Esamai FO. Health problems of street children in Eldoret, Kenya. East Afr Med J. 2001 Dec;78(12):624-9. doi: 10.4314/eamj.v78i12.8930. PMID 12199442
- [Background] Davey G, Tekola F, Newport MJ. Podoconiosis: non-infectious geochemical elephantiasis. Trans R Soc Trop Med Hyg. 2007 Dec;101(12):1175-80. doi: 10.1016/j.trstmh.2007.08.013. Epub 2007 Oct 31. PMID 17976670